CLINICAL TRIAL: NCT05982002
Title: Effect of Shock Wave Therapy on Truncal Obesity and Lipid Profile in Obese Post Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda mohammed fathey, Physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/002823
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Obesity
Keywords: Obesity-menopause-shock wave-lipid profile
MeSH Terms: conditions — Obesity | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Group A: (Control group)20 post menopausal women received moderate intensity aerobic exercise in addition to energy restricted diet 2time/week for 6 -weeks
  Interventions: Other: Moderate intensity aerobic exercise; Other: Energy-restricted diet
- Shock wave group (Experimental): Group B: (shock wave group)20 post menopausal women received the same intervention as in group A and 12 sessions of shockwave on abdomen twice/week for 6 -weeks
  Interventions: Device: shock wave; Other: Moderate intensity aerobic exercise; Other: Energy-restricted diet

INTERVENTIONS:
Device: shock wave — ESWT (Chattanooga, Intelect RPW, USA) continues mode, hand piece transmitter R SW D20 /20mm, with the following Parameter: Shock pressure of 3-4 bars, wave frequency of 12 Hz.
  Other Names: Extracorporeal shock wave therapy
  Arms: Shock wave group
Other: Moderate intensity aerobic exercise — Treadmail training exercise 60%-75% of Maximum heart rate MHR 2 times/ week
Other: Energy-restricted diet — energy intake was 500K calorie below daily requirements on average three meals at the same time of the day

SUMMARY:
This study aimed to evaluate the effect of six weeks extracorporeal shockwave therapy (SWT) on truncal obesity and serum lipids in obese postmenopausal women

DETAILED DESCRIPTION:
Truncal obesity occurs when the excess abdominal fat around the stomach and abdomen has accumulated to the point where it is likely to have a negative influence on health , increased visceral abdominal fat (VAF) is directly related to abdominal obesity (AO), which is also linked to endothelial dysfunction, inflammation, insulin resistance, diabetes mellitus, hypercholesterolemia, hepatic steatosis metabolic syndrome [MetS] and cancer.

High density lipoprotein (HDL) cholesterol, often known as cardio protective cholesterol, increases in a hypoestrogenic state such postmenopausal status, whereas triglyceride (TG), total cholesterol, and LDL cholesterol levels fall The prevention of CVD and dyslipidemia depends on the management of truncal obesity, and the reduction of serum lipid levels.

Extracorporeal shock wave therapy (ESWT) has lately been popular for treating fat-related disorders by altering the permeability of lipocyte membranes, improving blood flow and hastening macrophages' clearance of debris so cellulite, body contouring and localized fat can all be treated with the safe and non-invasive ESWT technology because to its mode of action in biological tissue In order to identify the best methods for treating abdominal obesity and prevent the risk of developing cardiovascular disease (CVD) in post-menopausal women. The current randomized controlled trial aimed to determine the effect of extracorporeal shockwave therapy (SWT) on truncal obesity and serum lipids in obese postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Obese Post menopausal women Body mass index more than or equal 30kg/m2 Waist circumference more than or equal 88 cm Waist hip ratio more than or equal 0.88cm Women not engaged in any procedure to treat obesity or received medication from 6 months

Exclusion Criteria:

* women diagnosed with malignancies or received chemical or radiotherapy or hormone replacement therapy or corticosteroids or diagnosed with liver disease or active infection or trauma

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Anrhropometric measurement | Before and after 6 weeks of treatment
  involving weight, height, waist circumference and hip circumference measured for each post-menopausal woman . The weight and height were measured using a weight-height scale without shoes and with a thin layer of clothes then calculate the body mass index according to the following equation: BMI=weight/height2 (Kg/m2), for both groups (A&B), waist circumference were measured pare skin from standing position using tape measure at the narrowest level between the costal margin and the iliac crest at the end of gentle expiration, and the hip circumference was measured at the widest level over the buttocks. Then, waist/hip ratio was calculated by dividing the waist by the hip circumference before and after treatment program for all women in both groups (A and B)
Lipid profile measurement | Before and after 6 weeks of treatment
  Fasting sample of venous blood was collected in the morning from each woman in both groups (A&B) from a vein on the inside of the elbow or the back of the hand after use of local antiseptic for the skin to prevent infection .Serum levels of the total cholesterol (TC), high-density lipoprotein (HDL), low-density lipoprotein (LDL) and triglycerides (TG) was measured by cobas 311 analyzer using a commercially available assay kit according to the manufacturer's instructions (Roche
  Diagnostics GmbH).

CONTACTS AND LOCATIONS:
Overall Officials: Hala Hanafy, Study Director — Professor of physical therapy for women's health; Marwa Hasanin, Study Director — Assistant professor of physical therapy for women's health; Hossam Hussien, Study Director — Professor of gynaecology and obstetrics
Locations (1):
- Faculty of physical therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Troia S, Moreira AM, Pisco D, Noites A, Vale AL, Carvalho P, Vilarinho R. Effect of shock wave therapy associated with aerobic exercise on cellulite: A randomized controlled trial. J Cosmet Dermatol. 2021 Jun;20(6):1732-1742. doi: 10.1111/jocd.13791. Epub 2020 Oct 26. PMID 33053245
- [Background] Zhang X, Ma Y. Global trends in research on extracorporeal shock wave therapy (ESWT) from 2000 to 2021. BMC Musculoskelet Disord. 2023 Apr 20;24(1):312. doi: 10.1186/s12891-023-06407-9. PMID 37081473